CLINICAL TRIAL: NCT00314457
Title: A Randomized, Double-blind Trial Comparing the Analgesic Efficacy and Side Effects of Continuous Intraarticular Infusion of Bupivacaine Versus Normal Saline in Patients Undergoing Knee and Shoulder Operations
Brief Title: Efficacy Study of Continuous Intraarticular Infusion in Patients Undergoing Arthroscopic Knee and Shoulder Operations
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Bupivacaine has recently been shown to inhibit osteoclast formation in vitro.
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Anesthesiology Associates, Ltd. (Other)
Responsible Party: Harshad Gurnaney, MBBS, The Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2005-5-4294
Record Dates: First submitted 2006-04-12; First posted 2006-04-14 (Estimated); Last update posted 2009-07-13 (Estimated); Status verified 2009-07

CONDITIONS: ACL Repair; Meniscectomy; Bankart Repair
Keywords: pain control; intra-articular pain control device; ACL repair; Bankart Repair
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Bupivacaine — Patients receive either normal saline or Bupivacaine in normal saline that infuses intraarticularly for 48 hours.

SUMMARY:
The aim of this study is to determine whether the continuous intraarticular infusion of local anesthetics in the postoperative period can improve analgesia and patients satisfaction after knee and shoulder arthroscopy.

DETAILED DESCRIPTION:
We propose to evaluate the long-term efficacy of the continuous intraarticular delivery of local anesthetics via a disposable, self-regulated DonJoy Pain Control infusion pump. Patients will be randomly assigned to receive either an intra-articular infusion of bupivacaine 0.125%, or saline delivered at a rate of 5 ml/hr for 48 hours by a DonJoy® Pain Control infusion pump. Patients will receive a femoral block (FNB) and a sciatic block (SNB) for knee arthroscopy or an interscalene block (INB) for shoulder arthroscopy prior to surgery. After the operation, patients will receive morphine via a Patient Controlled Analgesia (PCA) pump for pain control. The patient will be admitted overnight to a Care Unit, with the PCA discontinued at discharge or 24 hours, whichever is earlier. If clinically indicated, the PCA may be extended at the discretion of the pain team. Upon discharge and during the 48 hour study period the patient will receive oral oxycodone and acetaminophen. The patient and their family will remove the DonJoy® Pain Control infusion pump 48 hours after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 11 and 19 years old.
* Knee and shoulder arthroscopy procedures

Exclusion Criteria:

* Contraindications to Femoral-Interscalene Nerve Block
* Conditions that affect the proper evaluation of pain and side effects.
* Intake of NSAIDs or opioids in the 12 hours prior to the operation
* Allergy to study medications

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2005-08; Primary Completion 2007-02 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the total amount of opioids and other analgesic medications consumed in the recovery room and during the 48 hour study period (intravenous and oral). | 48 hour post operatively

SECONDARY OUTCOMES:
Secondary endpoints will include the incidence of side effects, such as nausea, vomiting, sedation and itching, pain scores at defined time periods and patients' satisfaction. | 48 hours post operatively

CONTACTS AND LOCATIONS:
Overall Officials: Harshad Gurnaney, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States